CLINICAL TRIAL: NCT01243632
Title: A Phase II Trial of Low-dose Gemcitabine in Prolonged Infusion and Cisplatin in Treatment of Malignant Pleural Mesothelioma
Brief Title: Gemcitabine in Long Infusion and Cisplatin for Malignant Pleural Mesothelioma Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: Ministry of Higher Education, Science and Technology, Solvenia (Other Government)
Responsible Party: Viljem Kovac, MD, Head of the Mesothelioma Team, Institute of Oncology Ljubljana
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 86/12/02
Record Dates: First submitted 2010-11-10; First posted 2010-11-18 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: malignant pleural mesothelioma; chemotherapy; gemcitabine; cisplatin; long infusion
MeSH Terms: conditions — Mesothelioma, Malignant

INTERVENTIONS:
Drug: Prolonged 6-hr infusion of gemcitabine — Gemcitabine 250 mg/m2 in prolonged 6 hr infusion on day 1 and 8, and cisplatin at 75 mg/m2 on day 2 of 3 week cycle, for 4-6 cycles

SUMMARY:
Combination of gemcitabine-cisplatin was one of the most effective chemotherapy treatment in mesothelioma patients. However, median survival of this patient group was only about 12 months. With intent to find more effective treatment the investigators performed phase II study with gemcitabine in low dose (130-250 mg/m2) in 6-hours (prolonged) infusion in combination with cisplatin in advanced non-small cell lung cancer (Zwitter et al. Anticancer Drugs 2005;16:1129-34). After favourable experience, the investigators decided to explore such regiment in patients with malignant pleural mesothelioma (MPM) as well.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate new regimen of treatment for its activity in malignant pleural mesothelioma (MPM). The primary objectives of the trial are assessing the treatment toxicity, response rate, and progress free survival; secondary objectives are assessment of overall survival and quality of life.

Inclusion criteria:

* Biopsy-proven diagnosis of MPM
* Inoperable for anatomic or physiological reason
* Measurable and previously unirradiated lesion
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 - 2
* Adequate haematopoietic, liver, and kidney function.
* Signed informed consent for participation in the trial

Exclusion criteria:

* Significant medical co-morbidity
* Pregnant or lactating women
* History of the cancer in the previous 10 years or breast cancer ever.

The general treatment schedule will be identical for all patients: gemcitabine in 6-hours infusion on days 1 and 8, and cisplatin at 75 mg/m2 on day 2 of a 3-weekly cycle with standard antiemetic treatment using metoclopramide, dexamethasone, aprepitant, and granisetron. After 4 cycles, patients not in progression and without serious toxicity continued with additional 2 cycles of monotherapy with gemcitabine in prolonged infusion.

National Cancer Institute Common Toxicity Criteria (NCI CTC), version 2.0 will be used for grading the toxicity. In the day of administration of the cytotoxic drug complete blood cell count and chemistry panel will be performed, and the treatment will be reduced or avoided in the event of bone marrow suppression or decline in renal clearance. In cases of Grade I (NCI CTC, vs. 2.0) neutropenia and/or thrombocytopenia, the dose of gemcitabine will be reduced to 75%; the drug will be omitted with Grade II or greater neutro/thrombocytopenia. Cisplatin will be omitted in cases of Grade ≥ II nephrotoxicity and/or grade III nausea or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of malignant pleural mesothelioma
* Inoperable for anatomic or physiological reason
* Measurable and previously unirradiated lesion
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 - 2
* Adequate haematopoietic, liver, and kidney function.
* Signed informed consent for participation in the trial

Exclusion Criteria:

* Significant medical co-morbidity
* Pregnant or lactating women
* History of the cancer in the previous 10 years or breast cancer ever.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2002-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Response rate | Computerized tomography (CT) measurement of disease will be performed after 2nd cycle of chemotherapy and at the end of the treatment
  Efficacy of the treatment will be measured by response rate (RR) and disease control rate (DCR) using modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria for assessment of response in malignant pleural mesothelioma

SECONDARY OUTCOMES:
Safety and tolerability | During the study
  Safety and tolerability will be assessed by monitoring the adverse events during treatment and follow-up phase and graded according the NCI Common Toxicity Criteria (CTC), version 2.0. Participants will be followed until death or 2 to 7 years (average 4.5 years).

CONTACTS AND LOCATIONS:
Overall Officials: Matjaz Zwitter, MD, PhD, Study Director — Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia